CLINICAL TRIAL: NCT07189676
Title: PLANETDIET: Sustainable Diets and Cardiometabolic Health: a Multi-omics Approach in a Randomized Controlled Trial (RCT)
Brief Title: Sustainable Diets and Cardiometabolic Health
Acronym: PlanetDiet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Novo Nordisk Foundation (NNF) (Unknown); Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Marta Guasch Ferre, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-25030722; Protocol code (Registry Identifier: 115994)
Record Dates: First submitted 2025-08-28; First posted 2025-09-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cardiometabolic Diseases
Keywords: metabolomics; proteomics; sustainable diets; cardiometabolic health; nordic diet; randomised controlled trial; cardiometabolic risk factors; planetary health diet
MeSH Terms: interventions — Nutrition Assessment; phosducin; Diet, Vegetarian; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Planetary health diet (PHD) (Experimental): Receiving PDH dietary advice, behavioral support, PHD food boxes, and group visits focused on dietary behavioural changes.
  Interventions: Behavioral: Dietary advice (PHD); Behavioral: Behavioural support PHD; Behavioral: Food boxes PHD; Behavioral: Group visits PHD
- Ovo-lacto-vegetarian diet (Experimental): Receiving ovo-lacto-vegetarian dietary advice, behavioral support, ovo-lacto-vegetarian food boxes, and group visits focused on dietary behavioural changes.
  Interventions: Behavioral: Dietary advice (Ovo-lacto-vegetarian diet); Behavioral: Behavioural support (Ovo-lacto-vegetarian diet); Behavioral: Food boxes (Ovo-lacto-vegetarian diet); Behavioral: Group visits (Ovo-lacto-vegetarian diet)
- Control group (habitual diet) (Other): Receiving dietary advice, minimum behavioral support, non-specific food boxes, and group visits focused on general research and health topics.
  Interventions: Behavioral: Dietary advice (control); Behavioral: Behavioral support (control); Behavioral: Food boxes (control); Behavioral: Group visits (control)

INTERVENTIONS:
Behavioral: Dietary advice (PHD) — It consists of a written document outlining the PHD diet recommendations. Participants will receive: 1) information about the PHD guidelines by EAT-Lancet (a high-quality plant-based diet with a low allowance of intake of eggs, dairy, chicken, and fish, but strictly avoiding red and processed meat) adapted to be nutritionally adequate and culturally accepted in Denmark, 2) a meal planner for their calorie demands (templates for 2000 kcal/day; 2500 kcal/day; and 3000 kcal/day), 3) guidance on alternatives for substituting meat when cooking at home or eating out, and 4) information on seasonal fruits and vegetables. The meal planner will specify the amounts of eggs, dairy, chicken, and fish that each participant should consume based on their total energy demands. The PHD dietary advice focuses on limiting certain food groups (without excluding them) based on their health and environmental impact.
  Other Names: EAT-Lancet recommendations; PHD
  Arms: Planetary health diet (PHD)
Behavioral: Dietary advice (Ovo-lacto-vegetarian diet) — It consists of a written document outlining the ovo-lacto-vegetarian diet guidelines. Participants will receive information to adhere to a stricter plant-based diet with an intake of eggs and dairy, but avoiding chicken, fish, and red and processed meat, and guidance on alternatives for substituting meat when cooking at home or eating out. Recommendations on food quantity or on consuming local and seasonal foods will not be given to pinpoint differences in the environmental aspect between interventions.
  Other Names: vegetarian diet
  Arms: Ovo-lacto-vegetarian diet
Behavioral: Dietary advice (control) — It consists of a written document outlining the general recommendations of a healthy diet (i.e. consumption of fruits and vegetables, decreasing the intake of sugar-sweetened beverages, etc.) without any specific advice on the consumption of animal products.
  Arms: Control group (habitual diet)
Behavioral: Behavioural support PHD — This component is designed to help participants adhere to the PHD through four individual and personalized dietary visits with a dietitian. Participants will also have access to a digital recipe collection in the study app. Recipes will be tagged by meal type and by season.
  Arms: Planetary health diet (PHD)
Behavioral: Food boxes PHD — Food boxes will be sent to participants' homes. PHD food boxes will include seasonal and local fruits and vegetables, whole grain products, legumes, nuts, and dairy or milk alternatives. If allergies or intolerances are identified, the food boxes will be modified to maintain safety and dietary compliance.
  Arms: Planetary health diet (PHD)
Behavioral: Group visits PHD — Group visits will provide support through nutritional education, social interaction, and peer learning, all focused on the dietary behavior changes required by the intervention. PHD group visits will cover topics such as PHD principles, and the related environmental and health outcomes.
  Arms: Planetary health diet (PHD)
Behavioral: Behavioural support (Ovo-lacto-vegetarian diet) — This component is designed to help participants adhere to the ovo-lacto-vegetarian through four individual and personalized dietary visits with a dietitian. Participants will also have access to a digital recipe collection in the study app. Recipes will be tagged by meal type.
  Arms: Ovo-lacto-vegetarian diet
Behavioral: Food boxes (Ovo-lacto-vegetarian diet) — Food boxes will be sent to participants' homes. Ovo-lacto-vegetarian food boxes will include fruits and vegetables, whole grains, legumes, nuts, soy-based products, eggs, and cheese. Local and seasonal aspects will not be taken into consideration. If allergies or intolerances are identified, the food boxes will be modified to maintain safety and dietary compliance.
  Arms: Ovo-lacto-vegetarian diet
Behavioral: Group visits (Ovo-lacto-vegetarian diet) — Group visits will provide support through nutritional education, social interaction, and peer learning, all focused on the dietary behavior changes required by the intervention. Ovo-lacto-vegetarian group visits will cover topics such as plant-based eating and nutritional adequacy.
  Arms: Ovo-lacto-vegetarian diet
Behavioral: Behavioral support (control) — Participants will attend four short individual dietary visits with a dietitian, where they will review the recorded dietary data. Participants of the control group will not have access a recipe collection or meal planner.
  Arms: Control group (habitual diet)
Behavioral: Food boxes (control) — Food boxes will be sent to participants' homes. Control food boxes will include fruits and vegetables, potato, nuts, cheese, animal protein products and canned food. Local and seasonal aspects will not be taken into consideration. If allergies or intolerances are identified, the food boxes will be modified to maintain safety.
  Arms: Control group (habitual diet)
Behavioral: Group visits (control) — Group visits will provide support through general health education, social interaction, and peer learning. Control group visits will cover topics such as the role and importance of controls in RCTs and general well-being.
  Arms: Control group (habitual diet)

SUMMARY:
This study aims to investigate the effects of sustainable diets on traditional and novel cardiometabolic risk factors.

The primary objective is:

• To test the effects of a sustainable diet on traditional cardiometabolic risk factors, specifically, a metabolic health score.

The secondary objectives are:

* To test the effects of sustainable diets on blood lipids, inflammatory markers, glucose markers, and anthropometric and body composition markers.
* To test the effect of sustainable diets on circulating metabolomic profiles.
* To test the effects of sustainable diets on circulating proteomic profiles.

Participants will receive dietary interventions of a sustainable health diet, namely the PHD diet (Planetary Health Diet), an ovo-lacto-vegetarian diet, or a habitual diet following general recommendations for a healthy diet without advice on consumption of animal products. The three-arm parallel RCT will involve adults (45-70 years old) at cardiovascular risk.

The primary hypothesis is that targeted interventions to adopt sustainable diets will have beneficial effects on cardiometabolic biomarkers, metabolomic, and proteomic profiles, compared to the habitual diet in individuals at cardiovascular risk.

DETAILED DESCRIPTION:
Background: To promote sustainable diets for planetary and human health, the EAT-Lancet Commission called for a global dietary transformation by 2050, advocating a dietary pattern shift to align food systems with environmental sustainability and human health. The Planetary Health Diet (PHD) promotes a plant-based approach, emphasizing the consumption of whole grains, fruits, vegetables, nuts, and legumes, and limited amounts of seafood and poultry, while discouraging excessive intake of red and processed meat, added sugar, refined grains, and starchy vegetables. Despite the promotion of the popular EAT-Lancet diet, there is no Randomized Controlled Trial (RCT) evaluating the impact of this pattern on established and novel cardiometabolic biomarkers. The trial design addresses the recognized lack of RCTs evaluating changes in multi-omic profiles by adhering to different dietary interventions; the lack of RCTs on sustainable diets that consider environmental aspects; and overcome limitations of potential reverse causation and other biases from observational studies.

Investigation plan: Participants will be randomized to receive advice on changes in the overall dietary pattern from specialized dietitians. Participants in the PHD diet group will be guided to follow the EAT-Lancet recommendations adapted to be nutritionally adequate and culturally acceptable in Denmark (a high-quality plant-based diet with a low allowance of intake of eggs, dairy, chicken, and fish, but strictly avoiding red and processed meat). Participants in the vegetarian diet group will be advised to adhere to a stricter plant-based diet with an intake of eggs and dairy but avoiding chicken, fish, and red and processed meat, and no recommendations on food quantity or the environment. The two interventions will be compared with the control group, where participants will follow their habitual diet without specific advice on the consumption of animal products. The present RCT is not a weight loss trial, thus no total calorie restriction will be advised, and physical activity will not be promoted. A maximum alcohol consumption limited to 100 grams/week for men and women drinkers will be allowed.

Dietary considerations: The comparisons will allow us to address the unanswered question of whether the inclusion of moderate amounts of animal-based products in the context of a climate-friendly diet is superior to a stricter vegetarian diet. Vegan diets were not considered because of the difficulty in adherence in European settings and the potential for micronutrient deficiencies. The higher between-group contrast, considering both health and environmental impact is expected to be found for PHD vs control group.

The study will include an information meeting, screening visit, baseline visit, two visits during the intervention (1 month and 3 months), and a final visit at 6 months. Additionally, two group visits (at 2 and 4 months) will be conducted. Outcome parameters (a metabolic health score and its components) will be measured using blood samples obtained at baseline, 3 months, and final visit. Urine samples will be collected for the research biobank at the baseline, 1 month, 3 months, and final visit. Fecal samples will be collected at baseline and the final visit. Participants will wear continuous glucose monitors (CGM) for 10 days at baseline and at the end of follow-up.

Participants will have access to a study app that will include a timeline of the study, study materials including dietary recommendations, meal planners and recipes according to the intervention group, and instructions for collecting biosamples. Participants will also use the app to respond to self-reported questionnaires. Food boxes containing targeted products for each intervention will be distributed to participants at baseline, 1 month, and 3 months.

Participants will attend two group visits (5-15 participants), where they will receive educational material, information about the science behind the trial and have the opportunity to share experiences with their peers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (males and females) between 45 and 70 years of age at the time of inclusion.
* Participants must have at least two metabolic alterations: 1) Waist Circumference (WC) >102 cm (males) or >88 cm (females); 2) self-reported medication for blood pressure or blood pressure >130/85 mmHg; 3) self-reported prediabetes or non-fasting plasma glucose 140-199 mg/dL (prediabetes); 4) self-reported lipid-lowering medication or diagnosis of impaired blood lipids (triglycerides: ≥ 150 mg/dL; and HDL: men: < 40 mg/dL and women: < 50 mg/dL).
* Participants are not institutionalized, able to read and provide consent before participation, and willing to attend in-person visits at the study site.
* Participants should have access to a smartphone and computer, or tablet and must be internet-literate.
* Understand Danish both in writing and when spoken.

Exclusion Criteria:

* Participants with any serious illness or history of cancer within the past 5 years (except adequately treated localized basal cell skin cancer or in situ uterine cervical cancer).
* Diagnosed with diabetes mellitus, CVD event (myocardial infarction, revascularization procedure, or stroke), or atrial fibrillation.
* Participants with diagnosed psychiatric conditions or cognitive impairment.
* Current smokers including all kinds of nicotine-containing products.
* BMI >35 kg/m2.
* Known or suspected abuse of alcohol or recreational drugs. Regular alcohol consumption exceeding the Danish national guidelines (i.e., more than 10 standard drinks per week or more than 4 drinks on any single day) will be excluded.
* Pregnancy or planning a pregnancy in the next year.
* Not willing to consume chicken and fish or not willing to make dietary changes related to the intervention.
* Participants with multiple food allergies that could hinder adherence to the intervention.
* Any other issue that makes the project responsible (PI or medical responsible) doubt the eligibility of the volunteer.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolic health score | Baseline, 3 and 6 months
  A metabolic health score that summarizes clinical biomarkers from main pathways associated with CVD: triglycerides, HDL-c, fasting plasma glucose, systolic and diastolic blood pressure, and high sensitive C-reactive protein (hs-CRP) (as a marker of inflammation). A Z-score will be calculated for each variable. HDL-cholesterol standardized values will be multiplied by -1 to be directly proportional to the cardiometabolic risk. The final score will be determined as the average of the individual component Z-scores. Thus, the metabolic health score is a continuous variable with a mean of 0 and a standard deviation of 1; higher scores indicate higher risk

SECONDARY OUTCOMES:
Changes in low-lipoprotein-cholesterol concentrations (LDL-c) | Baseline, 3 and 6 months
  Venous blood samples will be collected. LDL-c will be measured in fasting samples.
Changes in high-lipoprotein-cholesterol concentration (HDL-c) | Baseline, 3 and 6 months
  Venous blood samples will be collected. HDL-c will be measured in fasting samples.
Changes in triglycerides concentration | Baseline, 3 and 6 months
  Venous blood samples will be collected. Triglycerides will be measured in fasting samples.
Changes in Apoliprotein A1 (ApoA1) concentration | Baseline, 3 and 6 months
  Venous blood samples will be collected. ApoA1 will be measured in fasting samples.
Changes in Apoliprotein B (ApoB) concentration | Baseline, 3 and 6 months
  Venous blood samples will be collected. ApoB will be measured in fasting samples.
Changes in fasting glucose | Baseline, 3 and 6 months
  Fasting glucose will be measured in blood
Changes in insuline | Baseline, 3 and 6 months
  insulin levels will be measured in blood
Changes in HA1c | Baseline, 3 and 6 months
  Concentration levels of hemoglobin A1c will be measured in blood
Changes in continuous glucose monitor (CGM) measures | Baseline and 6 months
  CGM will be used to measure interstitial glucose in free-living conditions over 10 days.
Changes in high-sensitive C-reactive protein concentrations | Baseline, 3 and 6 months
  High-sensitive C-reactive protein concentration in fasting blood samples will be measured
Changes in Interleukin 6 (IL-6) concentrations | Baseline, 3 and 6 months
  Interleukin 6 concentration in fasting blood samples will be measured.
Changes in systolic blood pressure | Baseline, 3 and 6 months
  Measurements should be preceded by at least 5 minutes of rest in a quiet setting without distractions. Participants should be seated comfortably, with their arms resting and maintaining silence while the measurements are being taken. Two measures are taken, and the mean of the two measures is used. If there is a difference >5 mmHg between the two measurements, a third measure will be taken, and the two closer measurements will be used to calculate the mean.
Changes in distastolic blood pressure | Baseline, 3 and 6 months
  Measurements should be preceded by at least 5 minutes of rest in a quiet setting without distractions. Participants should be seated comfortably, with their arms resting and maintaining silence while the measurements are being taken. Two measures are taken, and the mean of the two measures is used. If there is a difference >5 mmHg between the two measurements, a third measure will be taken, and the two closer measurements will be used to calculate the mean.
Changes in heart rate | Baseline, 3 and 6 months
  Measurements should be preceded by at least 5 minutes of rest in a quiet setting without distractions. Participants should be seated comfortably, with their arms resting and maintaining silence while the measurements are being taken. Two measures are taken, and the mean of the two measures is used.
Changes in body weight | Baseline, 3 and 6 months
  Body weight (kg) will be measured with minimal clothing. The same calibrated equipment will be used for the respective measurements, and all study staff involved will be trained in handling the equipment and performing the measurements.
Changes in waist circumference | Baseline, 3 and 6 months
  The waist circumference will be measured using a flexible anthropometric tape (cm)
Changes in body mass index | Baseline, 3 and 6 months
  The body mass index will be calculated by dividing the weight (kg) by the square of height (m^2).
Changes in fat (%) | Baseline, 3 and 6 months
  Dual-energy X-ray Absorptiometry (DXA) scan will be performed in the morning in order to measure fat percentage (%). Participants are asked to meet fasting during the preceding 8 hours and to drink 400 mL of water before the measurement to ensure fluid balance.
Changes in lean mass | Baseline, 3 and 6 months
  Dual-energy X-ray Absorptiometry (DXA) scan will be performed in the morning in order to measure lean mass. Participants are asked to meet fasting during the preceding 8 hours and to drink 400 mL of water before the measurement to ensure fluid balance.
Changes in plasma metabolome | Baseline, 3 and 6 months
  Targeted metabolomics analysis will be conducted on plasma samples using a combination of liquid chromatography and high-resolution mass spectrometry. The concentration of 400 metabolites, including amino acids, acylcarnitines, tricarboxylic acid cycle metabolites, bile acids, purines, and pyrimidines will be measured.
Changes in plasma lipidome | Baseline, 3 and 6 months
  Targeted lipidomic analysis will also be carried out in plasma samples using liquid chromatography coupled with a trapped ion mobility spectroscopy time of flight mass spectrometer (LC-TIMS-TOF-MS). The concentration of 300 lipids will be annotated.
Changes in plasma proteome | Baseline, 3 and 6 months
  The Olink® Explore HT platform is a high-throughput, multiplex immunoassay platform intended to measure the relative concentration of proteins in liquid biopsies. The platform uses Olink's PEA™ technology coupled with a Next Generation Sequencing (NGS) readout method (NovaSeq6000 S4). The Olink® Explore HT analysis measures 5416 proteins using 2mL of sample volume with a specificity of 99.5% and negligible cross-reactivity. The outputted raw counts data is first processed using Olink® Explore Pre-processing software ngs2counts (version 4.5.0) and then quality-controlled using Olink® NPX Explore HT software (version 2.2.1) before generation of the Normalized Protein eXpression (NPX) values, Olink's unit of protein expression level in a log2 scale.

OTHER OUTCOMES:
Food biomarkers | Baseline, 1, 3 and 6 months
  The concentration of biomarkers characterizing specific food groups (e.g., red meat, fish) will be analyzed in urine samples by liquid chromatography-mass spectrometry, to assess compliance with the targeted food groups.
Dietary intake of key food groups | Baseline, 1, 3 and 6 months
  Intake of major food groups (eg., g/day of whole grains, legumes, fruits and vegetables, dairy foods) will be calculated. This information will come from 4-days dietary registries.
Dietary intake of key nutrients | Baseline, 1, 3 and 6 months
  Intake of saturated fatty acid, total fat, total sugars, fiber, and sodium intake will be calculated. This information will come from 4-days dietary registries.
Bone metabolism | Baseline, 3 and 6 months
  e.g., Concentration levels (ng/mL) of C-Terminal Telopeptide of Type I Collagen (CTX), Procollagen Type 1 N-Terminal Propeptide (P1NP)).
Changes in liver function | Baseline, 3 and 6 months
  concentration (U/L) of AST , ALT, GGT
Changes in kidney function | Baseline, 3 and 6 months
  concentration (mg/dL) of creatinine and uric acid
Changes in protein and albumin concentration | Baseline, 3 and 6 months
  concentration (g/L) of total proteins and albumin
Environmental footprint of the dietary interventions | Baseline, 1, 3 and 6 months
  Carbon dioxide equivalents of foods will be obtained using a carbon footprint database based on existing life cycle assessment data.
Dietary pattern acceptability | Baseline, 1, 3 and 6 months
  Participants will complete a Food Acceptability Questionnaire on the feasibility, acceptability, and satisfaction with the diet. A total of 8 questions with a 7-point response scales (1-7) will be asked.
Change in quality of life | Baseline, 1, 3 and 6 months
  Participants will complete the 12-item Short Form Health Survey (SF-12). Using the standard scoring algorithm, the Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) scores will be computed. Each summary score ranges from 0 to 100, with higher scores indicating better health outcomes.
Changes in 25-hydroxy-vitamin D3 concentration | Baseline, 3 and 6 months
  Vitamin D3 concentration will be measured.
Changes in vitamin B9 concentration | Baseline, 3 and 6 months
  Vitamin B9 concentration will be measured.
Changes in vitamin B12 concentration | Baseline, 3 and 6 months
  Vitamin B12 concentration will be measured.
Changes in ferritin concentration | Baseline, 3 and 6 months
  Ferritin concentration will be measured.
Changes in calcium concentration | Baseline, 3 and 6 months
  Calcium concentration will be measured.
Changes in cardiac function | Baseline, 3 and 6 months
  Measure of cardiac function throughout blood biomarker (e.g., Pro-B-type Natriuretic Peptide (proBNP))

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen. Rolighedsvej 26, DK-1958 Frederiksberg C., Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- See also: Related Info — https://eatforum.org/eat-lancet-commission/the-planetary-health-diet-and-you/